CLINICAL TRIAL: NCT06103045
Title: The Effects of Unilateral and Bilateral Mirror Therapy on Upper Extremity Function of Stroke at Acute Stage: A Pilot Randomized Controlled Trial.
Brief Title: The Effects of Unilateral and Bilateral Mirror Therapy on Upper Extremity Function of Stroke at Acute Stage.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111-168-E
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Stroke, Acute
Keywords: Stroke; unilateral mirror therapy; bilateral mirror therapy; acute stage; motor function of upper extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Patients with unilateral stroke and the onset within one month will be recruited and then randomly allocated to one of the three groups (including unilateral mirror therapy, bilateral mirror therapy, and conventional occupational therapy).
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors in charrge of pre- and post-test assessments were blinded to randomized allocation and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- unilateral mirror therapy (UMT) (Experimental): Participants will receive 30 minutes unilateral mirror therapy and then 30 minutes conventional occupational therapy in each treatment session. there will be 20 consecutive sessions (5 times per week, lasting 4 weeks totally)
  Interventions: Other: unilateral and bilateral mirror therapy
- Bilateral Mirror Therapy (BMT) (Experimental): Participants will receive 30 minutes bilateral mirror therapy and then 30 minutes conventional occupational therapy in each treatment session. there will be 20 consecutive sessions (5 times per week, lasting 4 weeks totally)
  Interventions: Other: unilateral and bilateral mirror therapy
- Conventional Occupational Therapy (COT) (Placebo Comparator): Participants will receive 60 minutes conventional occupational therapy in each treatment session. there will be 20 consecutive sessions (5 times per week, lasting 4 weeks totally)
  Interventions: Other: unilateral and bilateral mirror therapy

INTERVENTIONS:
Other: unilateral and bilateral mirror therapy — The mirror box is placed on a table in the sagittal plane of the participant. The affected upper extremity of the participant is hidden in the morror box and the unaffected upper extremity is placed symmetrically. During the unilateral or bilateral mirror therapy, the participant is requested to execute a serial of movements and tasks and pay attention on observing the reflection of the unaffected side in the mirror simultaneously. In the bilateral mirror therapy, the participant also has to move the affected upper extremity simultaneously; while in the unilateral mirror therapy, the participant only keeps the affected side relaxed.

SUMMARY:
Objective: To comparing the effects of unilateral and bilateral mirror therapy on upper extremity function of stroke at acute stage. We hypothesize there are different effects between unilateral and bilateral mirror therapy on stroke patients at acute stage. Method: Patients with unilateral stroke and the onset within one month will be recruited and then randomly allocated to one of the three groups (including unilateral mirror therapy, bilateral mirror therapy, and conventional occupational therapy). Patient will receive 20 consecutive sessions of intervention (5 time per week, totally 4 weeks) and assessments before and after the intervention within one week. In each intervention session, patients will receive 30 minutes unilateral or bilateral mirror therapy depending on their allocated groups and then 30 conventional occupational therapy. The patients recruited in the conventional occupational therapy group will receive 60 minute conventional therapy. The outcome measures at pre- and post-treatment will including the Fugl-Meyer Assessment for upper extremity (FMA-UE), the Modified Ashworth Scale (MAS), the Jamar Hydraulic Hand Dynamometer, the Chedoke Arm and Hand Activity Inventory (CAHAI), the Revised Nottingham Sensory Assessment (rNSA), and Functional Independence Measurement (FIM).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke onset within 1 month
* The score of Mini-Mental State Examination (MMSE) is more than 24
* The score of Fugl-Meyer Assessment for upper extremity (FMA-UE) is between 18 to 56
* The score of Modified Ashworth Scale (MAS) is less than 3
* Willing to receive 3-5 sessions of the intervention per week, total 20 sessions consecutively
* Willing to sign informed consent

Exclusion Criteria:

* Unstable vital sign or complicating with other symptoms of neurological disease
* Auditory or visual function impairment
* Complicating with perceptual impairment (e.g., apraxia, neglect, or visual agnosia)
* Receiving botulinum toxin injection within 3 months
* Complicating with Wernicke's or Broca's aphasia

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for upper extremity (FMA-UE) | pre-treatment: before intervention within a week; post-treatment: after intervention within a week
  The FMA-UE is a commonly used assessment in clinical for the extent of motor impairment of upper extremity post-stroke. The score ranged from 0 to 66. The psychometric properties of the FMA-UE had established, and there was also good responsiveness in the past studies.
The Jamar Hydraulic Hand Dynamometer | pre-treatment: before intervention within a week; post-treatment: after intervention within a week
  The Jamar Hydraulic Hand Dynamometer is a gold standard assessment tool for measuring muscle power including the grip strength, palmar pinch, and lateral pinch.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | pre-treatment: before intervention within a week; post-treatment: after intervention within a week
  The MAS is a clinical measurement for muscle spasticity. The score is ranged from 0 to 4. The shoulder, elbow, forearm, wrist, and fingers will be assessed. The psychometric properties of the MAS had established in the past studies.
Chedoke Arm and Hand Activity Inventory (CAHAI) | pre-treatment: before intervention within a week; post-treatment: after intervention within a week
  The CAHAI is used for the involvement of the impairment upper extremity during the bimanual tasks. There are 13 item and each score is ranged from 1-7. The psychometric properties of the CAHAI had established in the past studies.
Functional Independence Measurement (FIM) | pre-treatment: before intervention within a week; post-treatment: after intervention within a week
  The FIM was applied for evaluating the independent level and ADL function of the stroke patients. It includes 18 items of self-care, sphincter control, transfers, locomotion, communication, and social cognition. Score of each item is ranged from 1 to 7. The psychometric properties of the FIM had established in the past studies.
Revised Nottingham Sensory Assessment (rNSA) | pre-treatment: before intervention within a week; post-treatment: after intervention within a week
  The rNSA is developed for assessing sensory function of patients with stroke. The reliability of rNSA was established in the past study.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yi Lin, MS, Study Director — National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cauraugh JH, Summers JJ. Neural plasticity and bilateral movements: A rehabilitation approach for chronic stroke. Prog Neurobiol. 2005 Apr;75(5):309-20. doi: 10.1016/j.pneurobio.2005.04.001. PMID 15885874
- [Background] Geller D, Nilsen DM, Quinn L, Van Lew S, Bayona C, Gillen G. Home mirror therapy: a randomized controlled pilot study comparing unimanual and bimanual mirror therapy for improved arm and hand function post-stroke. Disabil Rehabil. 2022 Nov;44(22):6766-6774. doi: 10.1080/09638288.2021.1973121. Epub 2021 Sep 19. PMID 34538193
- [Background] Johnson D, Harris J, Stratford P, Richardson J. Inter-rater reliability of the Chedoke Arm and Hand Activity Inventory. NeuroRehabilitation. 2017;40(2):201-209. doi: 10.3233/NRE-161405. PMID 28222544
- [Background] Kidd D, Stewart G, Baldry J, Johnson J, Rossiter D, Petruckevitch A, Thompson AJ. The Functional Independence Measure: a comparative validity and reliability study. Disabil Rehabil. 1995 Jan;17(1):10-4. doi: 10.3109/09638289509166622. PMID 7858276
- [Background] Lee, M. T., Lu, Y. Y., Wu, C. Y., Hsieh, Y. W., & Lin, K.C. (2012). A systematic review of the effects of mirror therapy in patients with stroke. Journal of Taiwan Occupational Therapy Research and Practice, 8 (2), 125-140. doi:10.6534/jtotrp.2012.8(2).125
- [Background] Lincoln, N. B., Jackson, J. M., & Adams, S. A. (1998). Reliability and revision of the Nottingham Sensory Assessment for stroke patients. Physiotherapy, 84(8), 358- 365.
- [Background] Meseguer-Henarejos AB, Sanchez-Meca J, Lopez-Pina JA, Carles-Hernandez R. Inter- and intra-rater reliability of the Modified Ashworth Scale: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Aug;54(4):576-590. doi: 10.23736/S1973-9087.17.04796-7. Epub 2017 Sep 13. PMID 28901119
- [Background] Perez-Cruzado D, Merchan-Baeza JA, Gonzalez-Sanchez M, Cuesta-Vargas AI. Systematic review of mirror therapy compared with conventional rehabilitation in upper extremity function in stroke survivors. Aust Occup Ther J. 2017 Apr;64(2):91-112. doi: 10.1111/1440-1630.12342. Epub 2016 Dec 29. PMID 28032336
- [Background] Selles RW, Michielsen ME, Bussmann JB, Stam HJ, Hurkmans HL, Heijnen I, de Groot D, Ribbers GM. Effects of a mirror-induced visual illusion on a reaching task in stroke patients: implications for mirror therapy training. Neurorehabil Neural Repair. 2014 Sep;28(7):652-9. doi: 10.1177/1545968314521005. Epub 2014 Feb 18. PMID 24553103
- [Background] Zeng W, Guo Y, Wu G, Liu X, Fang Q. Mirror therapy for motor function of the upper extremity in patients with stroke: A meta-analysis. J Rehabil Med. 2018 Jan 10;50(1):8-15. doi: 10.2340/16501977-2287. PMID 29077129